CLINICAL TRIAL: NCT07001059
Title: oPtic Nerve Sheath Evaluation in gianT Cell aRtheritis by UltraSound
Acronym: PETRUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRD 0524; 2025-A00141-48 (Other: ANSM)
Record Dates: First submitted 2025-05-22; First posted 2025-06-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: Giant Cell Arteritis; Optic nerve sheath; Ultrasound
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orbital ultrasounds (Experimental): Orbital ultrasounds on patients suspected of GCA at the enrollment (M0) and at 6 months if the suspicion of GCA is confirmed after all the tests realized at the enrollment.
  Interventions: Diagnostic Test: orbital ultrasound

INTERVENTIONS:
Diagnostic Test: orbital ultrasound — orbital ultrasound at the beginning of the participation, and at 6 months after the inclusion.

SUMMARY:
The purpose of this study is to evaluate whether the measure of the optic nerve sheath is a reliable diagnostic marker for giant cell arteritis

DETAILED DESCRIPTION:
Giant Cell Arteritis (GCA) is a vasculitis affecting large and medium-sized vessels. It predominantly occurs in women, with a sex ratio of 3:1, and mainly affects individuals around 70 years of age. GCA is a rare condition, with an incidence of approximately 10 cases per 100,000 people in France.

Current recommendations suggest using imaging techniques and/or temporal artery biopsy (TAB) based on the clinical resources available. The key challenge in suspected cases of GCA is to establish a rapid diagnosis.

It is important to note that false-negative imaging results may occur if corticosteroid treatment is initiated prior to imaging: after 3 days for PET-CT, 5 to 7 days for Doppler ultrasound, and up to 14 days for TAB.

Diagnosing GCA is not always easy and depends on depends on the prompt performance of complementary examinations. Studies have shown that the optic nerve sheath is thickened on ultrasound in patients with GCA. In this context, the investigator aims to evaluate the measurement of the optic nerve sheath via ultrasound for diagnosing GCA. Ultrasound offers a faster, non-invasive, widely available, and cost-effective diagnostic tool.

ELIGIBILITY:
Inclusion Criteria:

* Patient with suspected GCA
* Patient over 50 years

Exclusion Criteria:

* Patient with history of GCA
* Patient with a history of polymyalgia rheumatic (PMR) without initial PET scan
* Patient with a history of retinal disease, demyelinating disease, or intracranial hypertension
* Use of corticosteroids > 0.5mg/kg in the last 2 weeks

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Assess whether the Optic Nerve Sheath Diameter (ONSD) measured by orbital ultrasound serves as an effective diagnostic marker for Giant Cell Arteritis (GCA) | At the patient enrollment visit and at 6 months
  Area under the ROC curve (AUC) of the optic nerve sheath measurements obtained by ultrasound during the enrollment phase, using the final clinical expert diagnosis at 6 months as the reference standard.
  The clinical expert's evaluation will be blinded to the optic nerve sheath measurements.

SECONDARY OUTCOMES:
Assess the reproducibility of the optic nerve sheath diameter (ONSD) measurements by ultrasound. | At the patient enrollment visit and at 6 months
  Mean bias according to Bland-Altman analysis, limits of agreement with their confidence intervals, maximum acceptable difference (clinical and statistical difference calculated using the root sum of squares of the coefficients of variation), inter-rater ICC.
Evaluate the diagnostic performance of ONSD in GCA. | At the patient enrollment visit and at 6 months
  Sensitivity, specificity, ROC curve inflection point (pathological threshold value), positive predictive value, negative predictive value, positive likelihood ratio, negative likelihood ratio.
Study the evolution of ONSD under treatment between M0 and M6 in patients with GCA. | At the patient enrollment visit and at 6 months
  Measurement of the optic nerve sheath diameter (ONSD) by ultrasound at baseline (within 3 days of corticosteroid initiation) in all patients, and at 6 months in patients with GCA.
Exploratory evaluation of ONSD according to the presence or absence of extracranial GCA. | At the patient enrollment visit and at 6 months
  Comparison of mean ONSD between subgroups: cranial GCA, extracranial GCA, and GCA-negative patients.
Exploratory evaluation of ONSD based on the presence or absence of GCA with visual involvement. | At the patient enrollment visit and at 6 months
  Comparison of mean ONSD between subgroups: GCA with visual involvement, GCA without visual involvement, and GCA-negative patients
Assess the feasibility of ultrasound as a diagnostic tool for GCA. | At the patient enrollment visit and at 6 months
  Description of the patient flow : average duration of the exam
Assess the feasibility of ultrasound as a diagnostic tool for GCA. | At the patient enrollment visit and at 6 months
  Description of the patient flow : percentage of exams performed, and percentage of interpretable exams.
Assess the feasibility of ultrasound as a diagnostic tool for GCA. | At the patient enrollment visit and at 6 months
  Description of the patient flow : number of exams performed, and number of interpretable exams.

CONTACTS AND LOCATIONS:
Overall Officials: Omar AL TABAA, Dr, Principal Investigator — Hôpital NOVO
Locations (9):
- France (9):
  - Rhumatology departement - Centre Hospitalier Aix en Provence, Aix-en-Provence
  - Rhumatology department - Centre Hospitalier Universitaire de Brest, Brest
  - Internal Medecine Department- CHU Caen, Caen
  - Internal Medicine and Clinical Immulogy department - Centre Hospitalier Universitaire de Dijon, Dijon
  - Internal Medicine and VascularMedecine Department - Centre Hospitalier Universitaire de Nantes, Nantes
  - Internal Medicine department - Hôpital Saint-Antoine, Paris
  - Rhumatology department - Hôpital Bichat, Paris
  - Rhumatology department - Hôpital NOVO - Pontoise site, Pontoise
  - Rhumatology department - Centre Hospitalier Universitaire de Tours, Tours